CLINICAL TRIAL: NCT00058864
Title: Trochanteric Padding to Prevent Hip Fractures
Brief Title: The HIP Impact Protection Program (HIP PRO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AG0001; 5R01AG018461-02 (NIH)
Record Dates: First submitted 2003-04-14; First posted 2003-04-15 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

INTERVENTIONS:
Device: Energy absorbing and distributing trochanteric pad

SUMMARY:
HIP PRO is a multicenter randomized, controlled trial of an energy absorbing and distributing padding system designed to reduce the incidence of hip fractures in 546 nursing home (NH) residents. The trial is being conducted in three geographic regions of the US: Boston, St. Louis, and Baltimore. Non bed- or chair-bound residents over the age of 65 are given protective underwear containing a single pocket and hip pad so that each resident becomes his/her own control. During the trial, hip fracture incidence will be compared in padded and unpadded hips using an intent to treat analysis. A secondary aim is to identify resident and facility factors contributing to non-adherence with the use of the hip protector.

DETAILED DESCRIPTION:
The HIP PRO Study is a randomized, controlled trial of the efficacy of a trochanteric padding system in the reduction of hip fractures in nursing home residents over the age of 65 in up to 45 nursing homes in three regions: Boston, MA, St. Louis, MO, and Baltimore, MD. Eligible residents of these facilities will be screened and then evaluated during a two week run-in period during which a hip protection compliance rate of at least 67% will be required for enrollment. Recruitment of all eligible residents entering each nursing home will continue throughout the 3.5 year follow-up period.

Each subject will be given a set of 4-6 protective underwear containing a single pocket and protective pad so that each resident becomes his/her own control. The side to be protected will be based on the randomization of nursing home facilities to either right or left-sided hip protection. The hip protection underwear is designed so that it may be worn during the day and while in bed at night. Several types of underwear have been designed for residents with special needs (e.g. incontinence, dementia). Compliance and efficacy are monitored at least three times weekly across all three nursing shifts.

A hip fracture adjudication committee, blinded to the side of the fracture, will review all information (including hospital records and radiologists' reports or hip radiographs) and issue a decision on whether a fracture has occurred. Primary analyses will be performed using an "intention to treat" approach. Secondary analyses will investigate resident and nursing home factors associated with hip protection compliance and effectiveness. An independent Data and Safety Monitoring Board (DSMB) has been convened and will review hip fracture rates and adverse event data at regular intervals.

Institutions participating in HIP PRO are: a Data Coordinating Center at Maryland Medical Research Institute in Baltimore, MD; three Clinical Centers at Washington University School of Medicine in St. Louis, MO, the University of Maryland in Baltimore, MD with the University of North Carolina in Chapel Hill, NC, and the Hebrew Rehabilitation Center for Aged in Boston, MA. The Data Coordinating Center will direct the overall administrative management of the trial.

ELIGIBILITY:
* Resident of eligible nursing home for at least two weeks
* Occupying a non-Medicare, non-acute, non-rehabilitation bed in the nursing home
* Over age 65
* Capable of independent transfer, not chair- or bed-bound
* Must give informed consent

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 546
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Maryland Medical Research Institute, Baltimore, Maryland
  - Hebrew Rehabilitation Center for Aged Research and Training Institute, Boston, Massachusetts
  - Washington University School of Medicine, Division of Geriatrics & Gerontology, St Louis, Missouri

REFERENCES:
- [Derived] Kiel DP, Magaziner J, Zimmerman S, Ball L, Barton BA, Brown KM, Stone JP, Dewkett D, Birge SJ. Efficacy of a hip protector to prevent hip fracture in nursing home residents: the HIP PRO randomized controlled trial. JAMA. 2007 Jul 25;298(4):413-22. doi: 10.1001/jama.298.4.413. PMID 17652295